CLINICAL TRIAL: NCT01646294
Title: An Exploratory Open Label, Three-way Crossover Study to Compare the Pharmacokinetic Profiles of Three Different YM178 Modified Release (OCAS) Formulations Under Fasted and Fed Conditions With YM178 Immediate Release (IR) Formulation Under Fasted Conditions in Healthy Subjects
Brief Title: A Study to Compare the Actions in the Body of Healthy Subjects of Three Modified Release Formulations of YM178 Under Fasted and Fed Conditions With One Immediate Release Formulation of YM178 Under Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 178-CL-030; 2004-003876-12 (EudraCT Number)
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Pharmacokinetics of YM178; Healthy Subjects
Keywords: Pharmacokinetics; Phase I; YM178; Modified release (Oral Controlled Absorption System (OCAS)); Immediate release (IR); Fasted conditions; Fed conditions
MeSH Terms: interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- OCAS-F (Experimental): YM178 OCAS tablet (OCAS-Fast) taken orally under fasted and fed condition
  Interventions: Drug: YM178 modified release (OCAS); Drug: YM178 immediate release (IR)
- OCAS-S (Experimental): YM178 OCAS tablet (OCAS-Slow) taken orally under fasted and fed condition
  Interventions: Drug: YM178 modified release (OCAS); Drug: YM178 immediate release (IR)
- OCAS-M (Experimental): YM178 OCAS tablet (OCAS-Medium) taken orally under fasted and fed condition
  Interventions: Drug: YM178 modified release (OCAS); Drug: YM178 immediate release (IR)

INTERVENTIONS:
Drug: YM178 modified release (OCAS) — oral
  Other Names: mirabegron; Myrebtriq
Drug: YM178 immediate release (IR) — oral
  Other Names: mirabegron; Myrebtriq

SUMMARY:
The purpose of the study is to investigate how quickly and to what extent YM178 is absorbed and eliminated from the body, and how well it is tolerated, when given in three different tablet formulations (sustained release) once a day with and without food, and to compare the results with the profile of the YM178 immediate release formulation taken twice daily without food.

DETAILED DESCRIPTION:
Subjects reside in the clinical research unit for 3 periods of 11 days each, with a washout period of at least 7 days between treatment periods. . Each subject is treated with multiple oral doses of the IR formulation (b.i.d.) under fasted conditions and, OCAS-F, OCAS-M or OCAS-S formulation (q.d.) under fasted and fed conditions (high fat breakfast).

The study is completed with a post-study visit between 7 and 14 days after discharge of period 3.

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 60.0 and 100.0 kg, and BMI between 18.0 and 30.0 kg/m2

Exclusion Criteria:

* Known or suspected hypersensitivity to β-adrenergic receptor agonists or constituents of the formulations used
* Clinically significant elevation of serum creatinine or liver enzymes as evidenced by creatinine and/or abnormal serum bilirubin
* Any clinically significant history of asthma, eczema, any other allergic condition or previous severe hypersensitivity to any drug
* Any clinically significant history of upper gastrointestinal symptoms in the 4 weeks prior to the first admission to the Research Unit
* Any clinically significant history of any other disease or disorder -gastrointestinal, cardiovascular, respiratory, renal, hepatic, neurological, dermatological, psychiatric or metabolic
* QTcB interval of >430 msec at screening (mean QTcB of two measurements>430msec)
* Abnormal pulse rate measurement (<40 or >90 bpm) at the pre-study visit after subject has been resting in supine position for 5 min
* Abnormal blood pressure measurements taken at the pre-study visit after subject has been resting in supine position for 5 minutes
* Positive orthostatic test at screening i.e. any symptoms of dizziness, light-headedness etc. and a fall of > 20 mmHg in systolic blood pressure after 2 min standing (as outlined in section 12.5) and an increase in pulse rate of ≥ 20 bpm
* History of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to first admission to the Research Unit.
* History of drinking more than 21 units of alcohol per week within 3 months prior to first admission to the Research Unit
* Donation of blood or blood products (more than 400 ml) within 3 months prior to first admission to the Research Unit or plasmapheresis within 4 weeks preceding the start of this study
* Positive serology test for HBsAg, HAV IgM, anti-HCV or anti-HIV 1+2
* Subject who is not willing to complete standard FDA high fat breakfast

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2005-01; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics profile of OCAS and IR assessed by plasma concentration | Day 1 & Day 6 - Day 8
  AUC0-12h (Area under the plasma concentration - time curve from t=0 to t=12h) Cmax (Maximum concentration), tmax (Time to attain Cmax) and Ctrough (Pre-dose plasma concentration)
Pharmacokinetics profile of OCAS assessed by plasma concentration | Day 8
  AUC0-24h (Area under the plasma concentration - time curve from t=0 to t=24h) Cmax, Tmax and Ctrough
Pharmacokinetics profile of IR assessed by plasma concentration | Day 8
  AUC0-12h , AUC12-24h (Area under the plasma concentration - time curve from t=12 to t=24h), AUC0-24h, PTR (Peak trough ratio), Cmax, Tmax and Ctrough

SECONDARY OUTCOMES:
Monitoring of safety parameters through assessment of vital signs, adverse events, Electrocardiogram (ECG) and clinical laboratory assessments | Baseline until Post Study Visit

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- Pharma Bio-Research B.V., Zuidlaren, Netherlands

REFERENCES:
- [Background] Lee J, Zhang W, Moy S, Kowalski D, Kerbusch V, van Gelderen M, Sawamoto T, Grunenberg N, Keirns J. Effects of food intake on the pharmacokinetic properties of mirabegron oral controlled-absorption system: a single-dose, randomized, crossover study in healthy adults. Clin Ther. 2013 Mar;35(3):333-41. doi: 10.1016/j.clinthera.2013.02.014. PMID 23497763